CLINICAL TRIAL: NCT01686295
Title: A Randomized, Double -Blind,, Sham-Device-Controlled, Multicenter, 24-Week Clinical Trial to Evaluate the Safety and Effectiveness of the iRestore ™ Hair Rejuvenation System in the Treatment of Male and Female Androgeneticalopecia
Brief Title: 24 Week Clinical Trial to Evaluate Safety and Effectiveness of a Hair Growth System to Treat Male and Female Baldness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Freedom Laser Therapy, Inc. (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CS940112; CS940112 (Other: FreedomLaser)
Record Dates: First submitted 2012-08-10; First posted 2012-09-18 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Androgenetic Alopecia
Keywords: androgenetic alopecia; Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- iRestore Hair Rejuvenation System (Experimental): Seventy six (76) subjects will be enrolled in the 24-week study; of which 38 will be male and 38 will be female using the iRestore hair growth device
  Interventions: Device: iRestore Hair Rejuvenation System
- Sham Device Arm (Sham Comparator): This study arm will use a sham device consistent with the experimental device with 12 men and 12 women with androgenetic alopecia 3 times a week for 30 minutes on non-consecutive days
  Interventions: Device: sham device

INTERVENTIONS:
Device: iRestore Hair Rejuvenation System — This study is to evaluate the effectiveness of the iRestore Hair Rejuvenation System when used as directed in promoting hair growth in men and women with androgenetic alopecia 3 times a week for 30 minutes on non-consecutive days
  Arms: iRestore Hair Rejuvenation System
Device: sham device — This shame device will be a sham comparator to evaluate the effectiveness of the iRestore Hair rejuvenation System when used as directed in promoting hair growth in men and women with androgenetic alopecia 3 times a week for 30 minutes on non-consecutive days
  Other Names: iRestore Hair Rejovenation System
  Arms: Sham Device Arm

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the iRestore Hair Rejuvenation System when used as directed in promoting hair growth in men and women with androgenetic alopecia

DETAILED DESCRIPTION:
The test treatment is the iRestore™ Hair Rejuvenation System. The device irradiates the scalp with visible light using 5 mW (class 3a) lasers. It is to be used approximately 3 times per week for approximately 30 minutes at each session.

The System is placed on the head and adjusted to a comfortable size by rotating knobs on the side of the device. If needed, subjects may replace the soft pad on the inside of the device with the thinner pad provided. There will be 2 options for using the product. The subject will either insert the 5-V AC power adapter pin into the device remote control, and the 5-V adapter will then be plugged into the AC outlet; or the subjects will use the rechargeable battery pack and belt clip. The battery pack is an external device which will allow the subject the freedom of mobility while treating the hair. The rechargeable battery pack will hold a charge for up to 3 hours prior to needing to be recharged. The iRestore™ remote control clips into the battery holster and the pack plugs into the remote. The battery pack can be placed in a pocket, clipped to the belt or placed next to the subject. The device will be turned on by pressing the power button on the remote control. The dome of the device is to be moved forward and backward by the subject to brush through the hair and increase the direct light which comes into contact with the scalp. Subjects will then position the dome at the front of the scalp and press the start button to begin a 10-minute session. Note: As a safety feature, the dome must be placed onto the head prior to starting the device. A timer will indicate the completion of the session with a beep sound. Subjects will complete the same process as done with the front of the scalp with the dome repositioned to the middle of the scalp and then the back of the scalp. Once all 3 positions have received the 10 minute treatment, the power button is to be held for approximately 3 seconds to turn the device off. Once off the device is to be unplugged from the wall.

The control device will be identical to the test device except that the laser-emitting units will be disabled. A standard light will be emitted from the device. Subjects and clinical staff engaged in the performance of assessments will be treatment blinded.

ELIGIBILITY:
Inclusion Criteria:

* Individuals eligible for inclusion in the study are those who:

  1. Are male or female, 25 to 60 years of age;
  2. If male, have Norwood-Hamilton classifications of IIa to V male pattern baldness;
  3. If female, have Ludwig Scale classifications I-4, II-1, II-2, or frontal;
  4. Are willing to have a tattoo created on the target area;
  5. Have been experiencing active hair loss within the last 12 months;
  6. In the case of females of childbearing potential, are using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom with spermicide, diaphragm with spermicide, abstinence or partner's vasectomy: abstinence or partner's vasectomy are acceptable if the female agrees to implement one of the other acceptable methods of birth control if her lifestyle or partner changes);
  7. Have Fitzpatrick Skin Type I-IV (See Table 1 Below);
  8. Are willing to have the target area hair clipped;
  9. Read, understand, and sign a photographic release form(s); and
  10. Read, understand, and sign an informed consent document after being advised of the nature of the study.

Table 1: Fitzpatrick Skin Types I Always burns easily, never tans II Always burns easily, tans minimally III Burns moderately, tans gradually (light brown) IV Burns minimally, always tans well (moderate brown) V Rarely burns, tans very well (moderate brown) VI Never burn, deeply pigmented

Exclusion Criteria:

* Individuals excluded from participation in the study are those who:

  1. Have used any of the following medications within 6 months prior to enrollment:

     * minoxidil, finasteride (or any other 5α-reductase inhibitor medications);
     * medications with anti-androgenic properties (eg, cyproterone, spironolactone, ketoconazole, flutamide, and bicalutamide);
     * topical estrogens, progesterone, tamoxifen, anabolic steroids;
     * medications that can potentially cause hypertrichosis (eg, ciclosporin, diazoxide, phenytoin, and psoralens);
     * oral glucocorticoids (inhaled glucocorticoids are permitted);
     * lithium or phenothiazines;
     * medications of known or suspected phototoxicity (eg, tetracyclines, thiazides, certain NSAIDs);
     * other medications which, in the opinion of the investigator, may interfere with the performance of study assessments or place the subject at undue risk;
  2. Will not agree to refrain from changing hair color and hair style during the course of the study;
  3. Have had a hair transplant, scalp reduction, hair weave, or tattoo which, in the opinion of the investigator, may interfere with the performance of the study assessments;
  4. Are using or have used depilatories, razors, or wax on the scalp to an extent which, in the opinion of the investigator, may interfere with the performance of the study assessments;
  5. Have psoriasis, active dermatitis/eczema, or severe acne on the scalp area;
  6. Have diabetes requiring exogenous insulin;
  7. Have cataracts;
  8. Have any medical condition which, in the opinion of the investigator, could affect hair growth (eg, Human Immunodeficiency Virus, connective tissue disease, inflammatory bowel disease);
  9. Have very little contrast between hair color and scalp, eg, are of a fair hair color (eg, white or very blond) and have very pale skin;
  10. Are females who are pregnant, planning to become pregnant during the study, or breastfeeding; and/or
  11. Are, in the opinion of the investigative personnel, unable to comprehend and/or otherwise comply with any aspect of study requirements.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-04 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Change from Screening/Baseline Hair Growth at Week 12 and Week 24 | Screening/Baseline, Week 12, and Week 24. The hair will be clean and properly combed for each individual in the following manner
  Standardized global scalp photographs will be taken of each subject prior to hair clipping for hair count macrophotography. These photographs will be obtained at Screening/Baseline, Week 12, and Week 24.To determine any differences from baseline photos.
  * Frontal (male only) and Top Scalp Views (female only): Hair will be center-parted and combed away from the part.
  * Vertex View (male only): Hair will be combed away from the center of the vertex like the spokes of a wheel.
  Global scalp photographs will be sent to Canfield Scientific, Inc. a central core lab for study imaging.

SECONDARY OUTCOMES:
Visual Scalp Assessment | At Baseline, Week 4, Week 12, and Week 24 subjects will have their scalp evaluated by the dermatologist or a trained designee
  At Baseline, Week 4, Week 12, and Week 24 subjects will have their scalp evaluated by the dermatologist or a trained designee for any sign of irritation or dermatologic conditions (eg, erythema, edema, dryness, scaling). The grading scale provided in Table 5 will be used to categorize each condition:
  Table 5: Visual Scalp Assessment Scale SCORE RESPONSE 0 None
  1. Mild
  2. Moderate
  3. Severe

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dosik, MD, Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Research Inc., Paramus, New Jersey, United States